CLINICAL TRIAL: NCT03210571
Title: Clinical Investigation of the eyeWatch Glaucoma Drainage Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rheon Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3007
Record Dates: First submitted 2017-07-01; First posted 2017-07-07 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eyeWatch device (Experimental)
  Interventions: Device: eyeWatch system

INTERVENTIONS:
Device: eyeWatch system — The eyeWatch device is composed of an AGDD, a control unit and a draining plate
  Other Names: Adjustable glaucoma drainage device (AGDD)

SUMMARY:
This study aims to test a new medical device, called the eyeWatch, used in filtering surgery for the treatment of glaucoma. This medical device has the following property: it allows better control of intraocular pressure in the initial postoperative phase by adjusting aqueous flow going through the device. The target criteria for the study are defined as: keeping intraocular pressure in target range; reducing the number of anti-glaucoma drugs; evaluating the number and type of postoperative complications. So far, this device has been already tested on 20 patients in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient shall suffer from primary open angle glaucoma, pseudo-exfoliative glaucoma, or refractory POAG or PEXG after previous failed filtering surgery, in the study eye. Diagnosis is based on glaucomatous optic neuropathy, Shaffer angle greater than 2 as seen on gonioscopy, and visual field defect attributed to glaucoma.
* Eye to be treated shall be phakic or pseudophakic with no other active ocular disease or disorder except for incipiens cataract. Prior ophthalmic surgery in the study eye shall have been performed more than 3 months before enrollment in this study.
* Patient condition is indicated for primary and secondary filtration surgery.
* Presence of elevated intraocular pressure defined as an intraocular corrected pressure (IOP) > 20 mmHg in the study eye, under maximally tolerated medications. The IOP level shall be obtained on 2 consecutive measurements (not taken on the same day) prior to surgery.
* Optic neuropathy is exclusively attributed to glaucoma.
* Patient agreed to sign the written inform consent prior to entering into the investigation.
* Patient is able and willing to complete post-operative follow-up requirements.

Exclusion Criteria:

* Diagnosis of neovascular glaucoma, congenital glaucoma.
* History of previous intraocular surgery in the study eye referring to but not limited to extraocular muscles (strabismus), corneal transplant, retinal surgery.
* Proliferative or severe non-proliferative retinopathy in either eye.
* Congenital anomaly of the anterior chamber angle in the study eye.
* Optic neuropathy other than glaucoma in the study eye.
* Patient with retinal vein occlusion in the study eye.
* Patient with retinal artery occlusion in the study eye.
* Patient with corneal opacifications, endotheliopathy, or irregularities that may interfere with the optic nerve evaluation or the IOP measurements in the study eye.
* Patient with a history of severe eye trauma in the study eye.
* Patient with ocular malformations such as microphthalmia in the study eye.
* Patient with concurrent inflammatory/infective eye disorder in the study eye.
* Patient with severe systemic disease or disabling conditions such as chronic renal failure, post organ transplants.
* Patient participating in another clinical trial or having participated in another clinical trial less than 3 months prior to entering into the investigation.
* Patient is pregnant, breast-feeding or unable to make the decision to participate in a clinical investigation (e.g. mentally ill person, mentally handicapped person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Number and type of serious adverse device events | Follow-up: day 1, Week 1, week 2, month 1, month 2, month 3, month 6, month 12 compared to baseline
  Demonstration of safety. The number and type of serious adverse device event per patient will be measured.
  Results of biomicroscopy, gonioscopy, pachymetry visual field and endothelial count will be compared to baseline.
Effectiveness in reducing the intraocular pressure | Follow-up: day 1, Week 1, week 2, month 1, month 2, month 3, month 6, month 12 compared to baseline
  Demonstration of the performance. The intraocular pressure (IOP in mmHg) will be measured at different time points to show the effective reduction compared to baseline. IOP reduced by ≥ 20% or IOP < 21 mmHg, and no IOP < 5 mmHg on two consecutive visits after 1 month (included)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan

REFERENCES:
- [Background] Villamarin A, Roy S, Bigler S, Stergiopulos N. A new adjustable glaucoma drainage device. Invest Ophthalmol Vis Sci. 2014 Mar 25;55(3):1848-52. doi: 10.1167/iovs.13-12626. PMID 24557347